CLINICAL TRIAL: NCT00855920
Title: A Multi-Center, Randomized, Double-Blind, Active-Controlled Study of the Safety and Efficacy of Rilonacept Administered Subcutaneously for the Treatment of an Acute Gout Flare
Brief Title: Study Utilizing Rilonacept in Gout Exacerbations
Acronym: SURGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IL1T-GA-0814
Record Dates: First submitted 2009-02-13; First posted 2009-03-05 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Acute Gout Flare
Keywords: Metabolism, Inborn Errors; Allopurinol; Metabolic Diseases; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Metabolic disorder; Purine-Pyrimidine Metabolism, Inborn Errors; Gout; Flare
MeSH Terms: conditions — Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Purine-Pyrimidine Metabolism, Inborn Errors; Gout | interventions — rilonacept; Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (for Rilonacept) and Indomethacin (Active Comparator): Two subcutaneous injections of Placebo (for Rilonacept) on Day 1 with Indomethacin orally thrice a day (TID) for 12 days (Indomethacin 50 mg for first 3 days and then, Indomethacin 25 mg for next 9 days).
  Interventions: Drug: Indomethacin; Other: Placebo (for Rilonacept)
- Rilonacept and Indomethacin (Active Comparator): Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) on Day 1 with Indomethacin orally TID for 12 days (Indomethacin 50 mg for first 3 days and then, Indomethacin 25 mg for next 9 days).
  Interventions: Drug: Rilonacept; Drug: Indomethacin
- Rilonacept and Placebo (for Indomethacin) (Active Comparator): Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) on Day 1 with Placebo (for Indomethacin) orally TID for 12 days.
  Interventions: Drug: Rilonacept; Other: Placebo (for Indomethacin)

INTERVENTIONS:
Drug: Rilonacept — Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) on Day 1 (Baseline).
  Arms: Rilonacept and Indomethacin; Rilonacept and Placebo (for Indomethacin)
Drug: Indomethacin — Indomethacin orally TID for 12 days (Indomethacin 50 mg for first 3 days and then, Indomethacin 25 mg for next 9 days).
  Arms: Placebo (for Rilonacept) and Indomethacin; Rilonacept and Indomethacin
Other: Placebo (for Indomethacin) — Placebo (for Indomethacin) orally TID for 12 days.
  Arms: Rilonacept and Placebo (for Indomethacin)
Other: Placebo (for Rilonacept) — Two subcutaneous injections of Placebo (for Rilonacept) on Day 1 (Baseline).
  Arms: Placebo (for Rilonacept) and Indomethacin

SUMMARY:
This purpose of this clinical research was to determine the efficacy and safety of an experimental drug called Rilonacept in participants with an acute gout attack. Participants participated in this study for 30 days. Rilonacept alone was being compared with Indomethacin alone and the combination of Rilonacept plus Indomethacin in treating acute gout flares.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 - 70 years of age
2. Previously met the preliminary criteria of ARA for the classification of the acute arthritis of primary gout
3. Presenting with an acute attack (flare) of gout within 48 hours of pain onset and pain of at least moderate severity
4. Must have at least 1 on the 0-3 scale for the swelling and the tenderness assessments of the gouty index joint
5. Current presentation of acute gout flare in 3 joints or less

Exclusion Criteria:

1. Treatment with any non-steroidal anti-inflammatory drug (NSAIDs) or opiates within 48 hours prior to baseline assessments. Treatment with long-acting NSAIDs within 1 month prior to baseline visit. Treatment with naproxen, meloxicam, nabumetone, celecoxib and indomethacin SR within 5 days prior to baseline visit.
2. Treatment with oral analgesics within 6 hours before baseline assessments. Treatment with topical analgesics within 12 hours before baseline assessments
3. History of NSAID intolerance
4. Participants with history of chronic, gouty arthritis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Evans, PharmD, Study Director — Regeneron Pharmaceuticals
Locations (43):
- United States (43):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Sierra Vista, Arizona
  - Burbank, California
  - Whittier, California
  - Clearwater, Florida
  - DeBary, Florida
  - DeLand, Florida
  - Jupiter, Florida
  - Orange Park, Florida
  - Orlando, Florida
  - Oviedo, Florida
  - Boise, Idaho
  - Elizabethtown, Kentucky
  - Baltimore, Maryland
  - Wheaton, Maryland
  - Detroit, Michigan
  - Stevenville, Michigan
  - Billings, Montana
  - Albuquerque, New Mexico
  - Albany, New York
  - Burlington, North Carolina
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Johnstown, Pennsylvania
  - Limerick, Pennsylvania
  - Norristown, Pennsylvania
  - Greenville, South Carolina
  - Bristol, Tennessee
  - Dallas, Texas
  - Forth Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - Mesquite, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Terkeltaub RA, Schumacher HR, Carter JD, Baraf HS, Evans RR, Wang J, King-Davis S, Weinstein SP. Rilonacept in the treatment of acute gouty arthritis: a randomized, controlled clinical trial using indomethacin as the active comparator. Arthritis Res Ther. 2013 Feb 1;15(1):R25. doi: 10.1186/ar4159. PMID 23375025
- See also: Rilonacept — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=501081761&QV1=RILONACEPT
- See also: Related Info — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?objectHandle=DBMaint&APPLICATION_NAME=drugportal&mergeData=true&actionHandle=default&nextPage=jsp%2Fdrugportal%2FResultScreen.jsp%3FprevPage%3Djsp%2Fdrugportal%2FChemidDataview.jsp%26OriginalSearc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 80 study sites in North America between 16 March 2009 and 26 February 2010. A total of 747 participants were screened in the study.
Pre-assignment Details: Out of 747 participants, 225 were randomized and treated in the study. Participants were randomized in 1:1:1 ratio to receive one of the three treatment groups (Placebo [for Rilonacept] + Indomethacin or Rilonacept 320 mg + Indomethacin or Rilonacept 320 mg + Placebo [for Indomethacin]) on Day 1 of the study.
Period: Overall Study
Arm/Group | Placebo (for Rilonacept) and Indomethacin | Rilonacept and Indomethacin | Rilonacept and Placebo (for Indomethacin)
Started | 76 | 74 | 75
Safety Population | 77 (1 participant from Rilonacept+Indomethacin arm received Placebo (for Rilonacept)+Indomethacin) | 73 (1 participant from Rilonacept+Indomethacin arm received Placebo (for Rilonacept)+Indomethacin) | 75
Completed | 68 | 65 | 64
Not Completed | 8 | 9 | 11
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lack of Efficacy | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Decision by the sponsor | 0 | 1 | 1
Not completed — Other than specified above | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included full analysis set (FAS) comprising of all randomized participants who received any study drug and had at least 1 post-baseline assessment.
Groups:
- Placebo (for Rilonacept) and Indomethacin: Two subcutaneous injections of Placebo (for Rilonacept) on Day 1 with Indomethacin orally TID for 12 days (Indomethacin 50 mg for first 3 days and then, Indomethacin 25 mg for next 9 days).
- Total: Total of all reporting groups
Arm/Group | Placebo (for Rilonacept) and Indomethacin | Rilonacept and Indomethacin | Rilonacept and Placebo (for Indomethacin) | Total
Number analyzed (Participants) | 75 | 74 | 73 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (10.90) | 48.6 (9.95) | 51.0 (10.83) | 50.3 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 13
  Male | 71 | 71 | 67 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 5 | 12
  Not Hispanic or Latino | 72 | 70 | 68 | 210
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 5 | 2 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 15 | 15 | 11 | 41
  White | 54 | 54 | 60 | 168
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient's Assessment of Pain Using a 5-Point Likert Scale (PAP-LS) in Index Joint to Averaged PAP-LS at 24, 48 and 72 Hours
Description: Participants were asked to complete a daily diary entry and assessed their pain in the past 24 hours using 5-point Likert Scale of 0 (None) to 4 (extreme pain), where; 0= none, 1= mild pain, 2= moderate pain, 3= severe pain, or 4= extreme pain. Change in PAP-LS in the index joint from baseline (Day 1) to the averaged PAP-LS values at 24, 48 and 72 hours was reported in this outcome measure (averaged PAP value= [PAP at 24 hours + PAP at 48 hours + PAP at 72 hours]/3).
Time Frame: Pre-dose on Day 1 (Baseline); post-dose at 4, 8, 12, 24, 48, 72 hours and then daily up to Day 13 or until gout flare ends
Population: Full analysis set (FAS) that included of all randomized participants who received any study drug and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Rilonacept) and Indomethacin | Rilonacept and Indomethacin | Rilonacept and Placebo (for Indomethacin)
Number analyzed (Participants) | 75 | 74 | 73
units on a scale | -1.40 (0.956) | -1.55 (0.919) | -0.69 (0.970)

2. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain Using a 5-Point Likert Scale (PAP-LS) in Index Joint at 72 Hours
Description: Participants were asked to complete a daily diary entry and assessed their pain in the past 24 hours using 5-point Likert Scale of 0 (None) to 4 (extreme pain), where; 0= none, 1= mild pain, 2= moderate pain, 3= severe pain, or 4= extreme pain.
Time Frame: Baseline (Day 1) to 72 hours
Population: Full analysis set (FAS) that included all randomized participants who received any study drug and had at least 1 post-baseline assessment. Here, number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Rilonacept) and Indomethacin | Rilonacept and Indomethacin | Rilonacept and Placebo (for Indomethacin)
Number analyzed (Participants) | 41 | 30 | 28
units on a scale | -1.41 (0.865) | -1.57 (1.104) | -1.29 (0.976)

3. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain Using a 5-Point Likert Scale (PAP-LS) in Index Joint at 48 Hours
Description: as for outcome 2
Time Frame: Baseline (Day 1) to 48 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Rilonacept) and Indomethacin | Rilonacept and Indomethacin | Rilonacept and Placebo (for Indomethacin)
Number analyzed (Participants) | 56 | 52 | 49
units on a scale | -1.36 (0.883) | -1.54 (0.959) | -1.08 (1.057)

4. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain Using a 5-Point Likert Scale (PAP-LS) in Index Joint at 24 Hours
Description: as for outcome 2
Time Frame: Baseline (Day 1) to 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (for Rilonacept) and Indomethacin | Rilonacept and Indomethacin | Rilonacept and Placebo (for Indomethacin)
Number analyzed (Participants) | 74 | 70 | 66
units on a scale | -1.16 (1.021) | -1.44 (0.895) | -0.55 (0.845)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Day 31) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the administration of dosing [Day 1] of study drug up to 35 days after the dose of study medication). Analysis was performed on safety population that included all participants who received any study drug and were analyzed according to the treatment actually received (as treated).
Groups:
- Placebo (for Rilonacept) and Indomethacin: Two subcutaneous injections of Placebo (for Rilonacept) on Day 1 with Indomethacin orally TID for 12 days (Indomethacin 50 mg for first 3 days and then, Indomethacin 25 mg for next 9 days). One participant randomized to treatment for Rilonacept and Indomethacin, received treatment for Placebo [for Rilonacept] and Indomethacin and analyzed in this arm.
- Rilonacept and Indomethacin: Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) on Day 1 with Indomethacin orally TID for 12 days (Indomethacin 50 mg for first 3 days and then, Indomethacin 25 mg for next 9 days). One participant randomized to treatment for Rilonacept and Indomethacin, received treatment for Placebo [for Rilonacept] and Indomethacin and analyzed in arm (Placebo [for Rilonacept] and Indomethacin).
Arm/Group | Placebo (for Rilonacept) and Indomethacin | Rilonacept and Indomethacin | Rilonacept and Placebo (for Indomethacin)
Serious Adverse Events (participants affected / at risk) | 0/77 | 3/73 | 0/75
Other Adverse Events (participants affected / at risk) | 8/77 | 7/73 | 7/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (for Rilonacept) and Indomethacin (N=77) | Rilonacept and Indomethacin (N=73) | Rilonacept and Placebo (for Indomethacin) (N=75)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (for Rilonacept) and Indomethacin (N=77) | Rilonacept and Indomethacin (N=73) | Rilonacept and Placebo (for Indomethacin) (N=75)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Institution will provide a copy of any publication to Sponsor prior to submission for review. Sponsor may request to remove confidential information from submission, provided that removal does not preclude the complete and accurate presentation and interpretation of the study results.